CLINICAL TRIAL: NCT06328595
Title: A Cross-Sectional Analysis of Muscular and Joint Symptoms in COVID-19 Patients: Insights From Syria
Brief Title: Muscular and Joint Symptoms in COVID-19 Patients: Insights From Syria
Status: Completed | Type: Observational
Sponsor: Syrian Private University (Other)
Responsible Party: Principal Investigator, Mohamad Zaid Mohamad Samer Ahmad Abdalla, Dr in Damascus university in general internal medicine, Syrian Private University
Other Study IDs: Cross sectional
Record Dates: First submitted 2024-03-22; First posted 2024-03-25 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Musculoskeletal Pain; COVID-19
Keywords: Fatigue; Joint pain; Covid-19 vaccination; Malaise
MeSH Terms: conditions — Musculoskeletal Pain; COVID-19; Fatigue; Arthralgia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Observation study, shows the relation between musckeloskeletal symptoms with during and post Covid-19 infection, by asking participants questions about there age,job,which vaccination covid participants took, residual area, social status, number of time of covid-19 infection, number of joint affected and duration of joint pain and asking if there any malaise or fatigue

ELIGIBILITY:
Inclusion Criteria:

* Participants aged ≥ 18 years with a prior COVID-19 infection or suspicious COVID-19 infection and currently residing in Damascus.

Exclusion Criteria:

* Participants below 18 years, those unwilling to give consent, individuals with joint surgery history, pregnant women, or those who had taken immunosuppressive drugs before the study.

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We collected participants by google form in syria
Sampling Method: Probability Sample
Enrollment: 1039 (Actual)
Dates: Start 2022-04-22 (Actual); Primary Completion 2023-05-04 (Actual); Study Completion 2023-08-20 (Actual)

PRIMARY OUTCOMES:
The Demographic characteristics were classified into four groups: Gender, Residual area, education level. | The study took 6 months to finish it with hard work, it was hard to reach our participants so we didn't only collect our data from google form we also colleted our data from Al-Mouassa University Hospital outpatients clinics and Damascus University
  Gender was either male or female. Residual area was divided into tow categories: Rural or City. Social status were divided into four types: Single, Married, Divorced, Widow .

CONTACTS AND LOCATIONS:
Locations (1):
- Mohamad Zaid Ahmad Abdalla, Damascus, Syria

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-24): https://cdn.clinicaltrials.gov/large-docs/95/NCT06328595/Prot_SAP_000.pdf